CLINICAL TRIAL: NCT01201655
Title: Multicentric Retrospective Case Control Study of the Impact of Hypersplenism and Splenectomy on Hepatocarcinogenesis in Patients With Posthepatitic Cirrhosis
Brief Title: Study of the Impact of Hypersplenism and Splenectomy on Hepatocarcinogenesis in Patients With Posthepatitic Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Air Force Military Medical University, China (Other); Xi'an Jiaotong University (Other)
Responsible Party: chen yong, Xijing Hospital
Other Study IDs: chenyong
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-01

CONDITIONS: Liver Cirrhosis; Carcinoma, Hepatocellular; Splenomegaly; Laparotomy
Keywords: Posthepatitic cirrhosis;; Hepatocarcinogenesis;; Splenectomy;
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular; Splenomegaly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate the impact of splenectomy coupled with portal-azygous disconnection on hepatocarcinogenesis in patients with post-hepatitic cirrhosis after hepatitis B or C virus infection by retrospective case-control study,We hope to find a new idear and method to prevent or cure HCC.

DETAILED DESCRIPTION:
A case-control study was carried out. The factors studied include age, gender, ascites, hepatic encephalopathy, ALT, AST, TBIL, ALP, GGT, Child-Pugh classification of liver function, and history of splenectomy with portal-azygous disconnection during the treatment of portal hypertension. According to the Child-Pugh classification, these cases were graded as A, B, and C. And according to the ranges of the normal reference values of the data, they were categorized into two groups including a normal group and an abnormal group.The data mainly comes from FMMU and Xi'an jiaotong university from the year of 2002 to 2012.

ELIGIBILITY:
Inclusion Criteria:

* after surgery

Exclusion Criteria:

* without surgery

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: post-hepatitic cirrhosis with portal hypertension and hypersplenism patients
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chen yong, professor, Study Director — Xia jielai
Locations (1):
- Chen yong, Xi'an, Shaanxi, China